CLINICAL TRIAL: NCT00002000
Title: A Study to Compare the Efficacy and Safety of Valacyclovir Hydrochloride ( 256U87 ) Versus Acyclovir in the Treatment of Recurrent Anogenital Herpes Infections in HIV Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 104A; 08
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Acyclovir; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Anus Diseases; Herpes Genitalis
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Anus Diseases; Herpes Genitalis | interventions — Valacyclovir; Acyclovir

INTERVENTIONS:
Drug: Valacyclovir hydrochloride
Drug: Acyclovir

SUMMARY:
To evaluate the safety and efficacy of oral valacyclovir hydrochloride (256U87) vs. acyclovir in the treatment of recurrent anogenital herpes in HIV-infected patients (CD4 greater than or equal to 100).

DETAILED DESCRIPTION:
Efficacy variables include the length of the episode, the time to lesion healing, the duration and severity of pain/discomfort, the duration of viral shedding, the proportion of patients with aborted episodes, the proportion of patients requiring extended therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* HIV-infected individual (CD4 = or > 100) with a history of recurrent anogenital herpes.
* Signed the consent form or present a signed parental consent form if below 18 years.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Hepatic impairments as evidenced by a three-fold increase from the upper limit of normal in alanine or aspartate transaminase. Impairment of renal function as evidenced by any elevation above the upper limit of normal for serum creatinine. History of hypersensitivity to acyclovir. Malabsorption or vomiting that would, in the investigators opinion, potentially limit the retention and absorption of oral therapy.

Patients with the following are excluded:

* Hepatic impairment as evidenced by a three-fold increase from the upper limit of normal in alanine or aspartate transaminase. Impairment of renal function as evidenced by any elevation above the upper limit of normal for serum creatinine.
* History of hypersensitivity to acyclovir. Malabsorption or vomiting that would, in the investigator's opinion, potentially limit the retention and absorption of oral therapy.

Prior Medication:

Excluded:

* Systemic antiherpes or immunomodulatory therapy within 30 days prior to entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Univ of South Alabama, Mobile, Alabama
  - ViRx Inc, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Denver Public Health Dept / Disease Control Services, Denver, Colorado
  - West Haven Veterans Administration Med Ctr, West Haven, Connecticut
  - Univ of South Florida, Tampa, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Northwestern Memorial Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Louisiana State Univ Med School, New Orleans, Louisiana
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Univ of New Mexico School of Medicine, Albuquerque, New Mexico
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Vanderbilt School of Medicine, Nashville, Tennessee
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington